CLINICAL TRIAL: NCT01253629
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate AFQ056 in Adult Patients With Fragile X Syndrome
Brief Title: Safety and Efficacy of AFQ056 in Adult Patients With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2212; 2009-013667-19 (EudraCT Number)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-03

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Martin-Bell Syndrome; Genetic Diseases; X-Linked
MeSH Terms: conditions — Fragile X Syndrome; Genetic Diseases, Inborn | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 25 mg bid AFQ056 (Experimental): 1 capsule of 25 mg and 1 capsule of placebo per intake
  Interventions: Drug: AFQ056
- 50 mg bid AFQ056 (Experimental): 2 capsules of 25 mg per intake
  Interventions: Drug: AFQ056
- 100 mg bid AFQ056 (Experimental): 1 capsule of 100 mg and 1 capsule of placebo per intake
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator): 2 capsules of placebo per intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056 — AFQ056, was provided as hard gelatin capsules, 25mg and 100 mg oral dosage strengths, identical in appearance were used
  Arms: 100 mg bid AFQ056; 25 mg bid AFQ056; 50 mg bid AFQ056
Drug: Placebo — Placebo medication identical in appearance to active medication was provided
  Arms: Placebo

SUMMARY:
This Phase IIb study is designed to assess whether 3 doses of AFQ056 are safe and effective in treating the behavioral symptoms of Fragile X Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fragile X Syndrome, who are at least moderately ill based on a Clinical Global Impression Severity score of at least 4 and have qualifying scores on the ABC-C and IQ test at Visit 1

Exclusion Criteria:

* Advanced, severe or unstable disease that may interfere with the study outcome evaluations
* Cancer within the past 5 years, other than localized skin cancer
* Current treatment with more than two psychoactive medications, excluding anti-epileptics
* History of severe self-injurious behavior

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in behavioral symptoms of Fragile X Syndrome using the Aberrant Behavior Checklist - Community (ABC-C) Total score in Stratum I | 12 weeks
  The ABC-C is a 58-item questionnaire that should have been completed as much as possible by the same rater. It is comprised of five subscales (irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity and inappropriate speech) plus the total score which ranks from 0 to 174 in patients who were fully methylated (FM)

SECONDARY OUTCOMES:
Change from baseline in behavioral symptoms of Fragile X Syndrome (FXS) using the ABC-C Total score in Stratum II | 12 weeks
  The ABC-C is a 58-item questionnaire that should have been completed as much as possible by the same rater. It is comprised of five subscales (irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity and inappropriate speech). Assessing the reduction in the (ABC-C) total score after 12 weeks of treatment in FXS patients with partially methylated (PM) FMR1 gene.
Global improvement of symptoms in Fragile X using the Clinical Global Impression-Improvement (CGI-I) scale | 12 weeks
  The CGI-I score ranges from 1 to 7 (with 1 being "very much improved", 4 being "no change" to 7 being "very much worse")
Change from baseline in irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity, and inappropriate speech assessed by the individual subscales of the ABC-C scale | 12 weeks
  comprised of five subscales (irritability, lethargy/social withdrawal, stereotypic behavior, hyperactivity and inappropriate speech) plus the total score which ranks from 0 to 174
The proportion of patients with clinical response in the ABC-C total score | 12 weeks
  response is defined as reduction of at least 25% from baseline in the ABC-CFX total score and a score of 1 (very much improved) or 2 (much improved) on the CGI-I scale at Week 12
improvement of repetitive behavior as measured by changes in the RBS-R | Week 12
  The Repetitive Behavior Scale - Revised (RBS-R) includes six domains: ritualistic behavior, sameness behavior, stereotypic behavior, self-injurious behavior, compulsive behavior, and restricted interests. A negative change from baseline indicates improvement

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (12):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, Media, Pennsylvania
  - Novartis Investigative Site, Greenwood, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Australia (3):
  - Novartis Investigative Site, Ryde, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Caulfield, Victoria
- Canada (2):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Sherbrooke, Quebec
- Novartis Investigative Site, Glostrup Municipality, Denmark
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma, RM
- Spain (2):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Berry-Kravis E, Des Portes V, Hagerman R, Jacquemont S, Charles P, Visootsak J, Brinkman M, Rerat K, Koumaras B, Zhu L, Barth GM, Jaecklin T, Apostol G, von Raison F. Mavoglurant in fragile X syndrome: Results of two randomized, double-blind, placebo-controlled trials. Sci Transl Med. 2016 Jan 13;8(321):321ra5. doi: 10.1126/scitranslmed.aab4109. PMID 26764156
- See also: Results for CAFQ056A2212 from the Novartis Clinical Trial website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12423